CLINICAL TRIAL: NCT03509909
Title: Mechanisms of Change in Yoga and Physical Activity for Veterans
Brief Title: Yoga and Physical Activity for Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBB-007-17F; CX001647-01A1 (Other Grant/Funding Number: VA CSR&D)
Record Dates: First submitted 2018-04-17; First posted 2018-04-26 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: PTSD
Keywords: yoga; exercise; randomized controlled trial
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Motor Activity

STUDY DESIGN:
Intervention Model Description: Experimental condition: Manualized hatha yoga, a 12-session group-based yoga class led by a trained teacher Control condition: Manualized supportive physical activity, a 12-session group-based stretching and strengthening class led by a trained instructor
Who Masked: Outcomes Assessor
Masking Description: The outcome evaluator is blind to experimental condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hatha yoga (Experimental): 12- week group-based yoga class
  Interventions: Behavioral: Hatha yoga
- Supportive exercise (Active Comparator): 12-week group-based stretching and strengthening class
  Interventions: Behavioral: Supportive physical activity

INTERVENTIONS:
Behavioral: Hatha yoga — Manualized hatha yoga
  Arms: Hatha yoga
Behavioral: Supportive physical activity — Manualized stretching and strengthening
  Arms: Supportive exercise

SUMMARY:
Posttraumatic stress disorder (PTSD) is a major health problem for the nation's Veterans, leading to significant physical and mental health morbidity and mortality. Current empirically-supported interventions ameliorate symptoms but generally do not restore full functioning, so the development of alternative or complementary approaches is a critical need. Large numbers of Veterans are seeking out yoga as a part of their recovery plans, but there is not enough evidence to recommend yoga for treatment of PTSD. Likely reflecting this heterogeneity, evidence of yoga's efficacy is highly variable. This project aims to address this problem by comparing the effect of yoga to a matched exercise control condition. The study will also explore the mechanisms by which yoga impacts PTSD. Ultimately, the goal of this research would be to contribute to integrative care planning, whereby multiple approaches can be applied in a synergistic manner to restore wellness for Veterans affected by PTSD.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a chronic, debilitating condition with a broad negative impact on physical and mental health functioning. Excellent, empirically-supported interventions for PTSD are readily available to Veterans, but the majority of patients who receive the best available treatments continue to have a diagnosable disorder after treatment. This suggests that complementary interventions may be useful to fully restore functioning. In addition, many patients seek alternatives to psychotherapy or pharmacotherapy. This is evident in the increasing numbers of individuals with PTSD are turning to alternative approaches. At present, however, the investigators lack a good evidence base from which to make recommendations about the use of complementary and alternative approaches.

Yoga is very popular practice, touted to enhance physical, mental and spiritual well-being. Many Veterans with PTSD have turned to yoga as a part of their recovery plan, often seeking care outside the specialty mental health system. Initial evidence suggests that the practice leads to clinically significant change in symptoms, but results are yet inconclusive, particularly in Veterans. Thus, this project will provide additional data as to efficacy of yoga for Veterans PTSD.

The study is a randomized controlled trial involving approximately 100 Veterans with PTSD from the San Diego area. These Veterans will be randomized to receive a manualized hatha yoga intervention or a supportive exercise control condition. Both interventions will be delivered by trained instructors via livestreaming or recorded classes over a 12-week period. Assessment of clinical outcomes and methodological variables will take place before, during, immediately after, and 3-months after the intervention. Analyses will focus on change in the intervention groups over time and the degree to which change is associated with the candidate mechanisms.

Results of this study have the potential to inform the way in which yoga is delivered to Veterans as well as to increase knowledge about the underlying processes by which PTSD can be ameliorated. Given the high demand for yoga demand by individuals with PTSD and the degree to which the practice is already being provided in many clinical settings, findings from this study will be immediately relevant. Findings may also guide future research in complementary and alternative approaches by demonstrating the principle of targeting different processes of change to create an integrative care plan.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who have clinically meaningful PTSD symptoms

Exclusion Criteria:

* serious suicidality or homicidality that has required urgent or emergent evaluation or treatment within the past three months
* a known, untreated substance abuse or dependence problem

  * inclusion is possible if there is evidence that the individual has been afforded and is complying with treatment for the substance problem
* serious mental disorders, such as psychotic disorders or bipolar type I, or serious dissociative symptoms
* cognitive impairment that would interfere with treatment
* circumstances that lead to recurrent traumatization

  * e.g., engaged in a violent relationship
* any medical condition for which exercise is contraindicated, including pregnancy
* concurrent enrollment in any other treatment specifically targeting PTSD symptoms or in any meditative or mind-body intervention

  * including yoga practice >1 class/month in the preceding 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ariel J. Lang, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Specific parameters of sharing are not yet established

REFERENCES:
- [Background] Lang AJ, Malaktaris A, Maluf KS, Kangas J, Sindel S, Herbert M, Bomyea J, Simmons AN, Weaver J, Velez D, Liu L. A randomized controlled trial of yoga vs nonaerobic exercise for veterans with PTSD: Understanding efficacy, mechanisms of change, and mode of delivery. Contemp Clin Trials Commun. 2021 Jan 28;21:100719. doi: 10.1016/j.conctc.2021.100719. eCollection 2021 Mar. PMID 33604485

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hatha Yoga | Supportive Exercise
Started | 67 | 50
Completed | 46 | 37
Not Completed | 21 | 13
Not completed — Withdrawal by Subject | 16 | 9
Not completed — Lost to Follow-up | 3 | 4
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hatha Yoga | Supportive Exercise | Total
Number analyzed (Participants) | 67 | 50 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (13.2) | 48.4 (13.0) | 47 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 17 | 41
  Male | 43 | 33 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 9 | 30
  Not Hispanic or Latino | 44 | 41 | 85
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 3 | 5
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 8 | 15 | 23
  White | 39 | 26 | 65
  More than one race | 12 | 4 | 16
  Unknown or Not Reported | 1 | 0 | 1
Martial status [Count of Participants; unit: Participants]
  Divorced, separated or widowed | 16 | 11 | 27
  Married, common law or permanent partner | 37 | 31 | 68
  Never married | 14 | 8 | 22
Education [Count of Participants; unit: Participants]
  High school or GED | 16 | 10 | 26
  Some college | 21 | 17 | 38
  College degree | 12 | 11 | 23
  Post-college | 18 | 12 | 30
Employment [Count of Participants; unit: Participants]
  Full time | 28 | 17 | 45
  Not in paid workforce | 22 | 18 | 40
  Part time | 8 | 5 | 13
  Unemployed | 9 | 10 | 19

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale for Diagnostic and Statistical Manual Version 5 (CAPS-5)
Description: Semi-structured clinical interview assessing severity of PTSD symptoms administered by a trained, blinded assessor. The range of scores is 0-80. Mpre-Mpost is presented, so positive numbers indicate a reduction in PTSD symptom severity from before to after the intervention.
Time Frame: Baseline to post-treatment (approx 12 weeks)
Population: Differs from the total population due to missing data. Includes individuals with both time points because of the nature of the change score.
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Hatha Yoga | Supportive Exercise
Number analyzed (Participants) | 48 | 39
change in units on a scale | 3.92 (10.05) | 3.46 (10.55)
Statistical Analysis 1: Comparison: Hatha Yoga vs Supportive Exercise; Test type: Superiority; p = 0.74, Mixed Models Analysis

2. Secondary Outcome: Patient Health Questionnaire Depression Items (PHQ-9)
Description: Self-report measure of depressive symptoms with a range of 0-27. Mpre-Mpost is presented, so positive numbers indicate a reduction in depression severity.
Time Frame: Baseline to post-treatment (approx 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Hatha Yoga | Supportive Exercise
Number analyzed (Participants) | 43 | 36
change in units on a scale | 3.79 (6.01) | 2.11 (4.47)

3. Secondary Outcome: State-Trait Anxiety Inventory, State Subscale
Description: Self-report measure of anxiety symptoms with "state" and "trait" subscales; state is reported. The subscale scores range from 20 to 80. Mpre-Mpost is presented, so positive numbers indicate a reduction in anxiety.
Time Frame: Baseline to post-treatment (approx 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Hatha Yoga | Supportive Exercise
Number analyzed (Participants) | 44 | 32
change in units on a scale | 0.23 (5.61) | -0.53 (6.9)

4. Secondary Outcome: State-Trait Anger Expression Inventory - II (STAXI-II), State Anger Subscale
Description: Self-report measure of anger with three major subscales (state anger, trait anger and anger control index), which are quantified as T-scores (i.e., 50 indicates the population mean with a standard deviation of 10), calculated from published adult norms tables. Change in T-scores, Tpre-Tpost, is presented, so positive numbers indicate a reduction in anger.
Time Frame: Baseline to post-treatment (approx 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in T-score
Arm/Group | Hatha Yoga | Supportive Exercise
Number analyzed (Participants) | 46 | 36
change in T-score | 1.02 (9.65) | 1.08 (6.94)

5. Secondary Outcome: Insomnia Severity Index
Description: Self-report measure of insomnia with a range of 0-28. Mpre-Mpost is presented, so positive numbers indicate a reduction in sleep disturbance.
Time Frame: Baseline to post-treatment (approx 12 weeks)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: change in units on a scale
Arm/Group | Hatha Yoga | Supportive Exercise
Number analyzed (Participants) | 45 | 33
change in units on a scale | 2.73 (4.24) | 1.64 (4.94)

6. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference 4a
Description: Self-report measure of pain interference, reported as a T-score (i.e., 50 indicates the population mean with a standard deviation of 10) calculated from published adult norms table. Change in T-scores, Tpre-Tpost, is presented, so positive numbers indicate a reduction in pain interference.
Time Frame: Baseline to post-treatment (approx 12 weeks)
Population: Differs from the total population due to missing data. Includes individuals with both time points because of the nature of the change score. Loss of data increased as scale is invalid if all items are not answered.
Measure: Mean (Standard Deviation); unit: change in T-score
Arm/Group | Hatha Yoga | Supportive Exercise
Number analyzed (Participants) | 30 | 25
change in T-score | 0.8 (8.47) | 0.92 (6.05)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Hatha Yoga | Supportive Exercise
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/50
Serious Adverse Events (participants affected / at risk) | 2/67 | 1/50
Other Adverse Events (participants affected / at risk) | 25/67 | 29/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hatha Yoga (N=67) | Supportive Exercise (N=50)
Broken bones (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Acute injury secondary to a car accident
Alcohol withdrawal (Psychiatric disorders) | 1 (1) | 0 (0)
Overdose (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hatha Yoga (N=67) | Supportive Exercise (N=50)
Gastrointestinal issues (Gastrointestinal disorders) | 2 (2) | 5 (5)
Muscle/tissue soreness (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 9 (9)
Emotional distress (Psychiatric disorders) | 6 (6) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 4 (4)
Symptoms of illness, including cold, flu and COVID-19 (Infections and infestations) | 11 (11) | 8 (8)
Joint pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-16): https://cdn.clinicaltrials.gov/large-docs/09/NCT03509909/Prot_SAP_000.pdf